CLINICAL TRIAL: NCT02975557
Title: A Phase I/II Randomized, Placebo-Controlled, Double-Blind, Single-Center, Tolerability And Preliminary Efficacy Study Of Use of Brimonidine Eye Drops for Treatment of Ocular Graft-vs-Host Disease (oGVHD)
Brief Title: Brimonidine Eye Drops for Treatment of Ocular Graft-vs-Host Disease (oGVHD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual of subjects. May take longer than expected to complete the trial.
Sponsor: Sandeep Jain, MD (Other)
Collaborators: Ocugen (Industry)
Responsible Party: Sponsor-Investigator, Sandeep Jain, MD, Professor of Ophthalmology, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-0278
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Dry Eye; Ocular Graft vs Host Disease; Meibomian Gland Dysfunction
Keywords: Brimonidine; Dry Eye; oGVHD; MGD
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Brimonidine Tartrate; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brimonidine 0.15% (Active Comparator): Brimonidine 0.15% eye drops 2 times a day for 12 weeks
  Interventions: Drug: Brimonidine 0.15%
- Brimonidine 0.075% (Active Comparator): Brimonidine 0.075% (1:1 dilution will be performed using 0.15% Alphagan-P solution with Refresh Plus Artificial Tears solution) eye drops 2 times a day for 12 weeks.
  Interventions: Drug: Brimonidine 0.075%
- Placebo (Placebo Comparator): Placebo (Refresh plus Artificial Tear) dispensed in Brimonidine bottles 2 times a day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brimonidine 0.15% — Brimonidine 0.15% eye drops 2 times a day for 12 weeks
  Other Names: Alphagan P
  Arms: Brimonidine 0.15%
Drug: Brimonidine 0.075% — Brimonidine 0.075% (1:1 dilution will be performed using 0.15% Alphagan-P solution with Refresh Plus Artificial Tears solution) eye drops 2 times a day for 12 weeks.
  Other Names: Alphagan P
  Arms: Brimonidine 0.075%
Drug: Placebo — Placebo (Refresh plus Artificial Tear) dispensed in Brimonidine bottles 2 times a day for 12 weeks.
  Other Names: Refresh plus Artificial Tear
  Arms: Placebo

SUMMARY:
The objective of this study is to establish whether patients with dry eye disease (DED) are able to tolerate receiving Brimonidine: 0.15% eye drops two times a day for twelve weeks (primary tolerability objective) and to investigate the preliminary efficacy of Brimonidine 0.15% topical eye drop solution in treating Meibomian Gland Dysfunction (MGD) (primary efficacy objective).

Meibomian Gland dysfunction can happen with numerous conditions such as Rosacea, Sjögren's syndrome, and oGVHD. In order to limit the influence of differing etiologies on the outcome of this trial, the investigator has limited the screening to MGD that accompanies oGVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Capable of giving informed consent and does provide informed consent.
3. Diagnosis of Meibomian Gland Disease
4. Women must be post-menopausal ≥ 1 year, or surgically sterilized. If not, a negative urine pregnancy test is required within 7 days of the participant receiving first dose of study drug along with definite evidence of contraceptive use during the duration of the study. Women of reproductive age should use a method of birth control that is acceptable to the participant and the study doctor. This may include oral contraceptive pills, birth control implants, barrier methods or abstinence. If a participant suspects pregnancy after being enrolled, another pregnancy test will be administered. If the test is positive, the participant will be discontinued from the study immediately.

Exclusion Criteria:

1. Allergic to Brimonidine or any similar products, or excipients of Brimonidine
2. Currently receiving any Brimonidine preparation as a part of glaucoma management
3. Receiving or have received within 30 days any experimental systemic medication.
4. Active ocular infection or ocular allergies.
5. Any history of eyelid surgery or ocular surgery within the past 3 months.
6. Corneal epithelial defect larger than 1 mm2 in either eye.
7. Have active drug/alcohol dependence or abuse history.
8. Vulnerable populations, such as neonates, pregnant women, children, prisoners, institutionalized individuals, or others who may be considered vulnerable populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Jain, MD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Illinois Eye and Ear Infirmary, University of Illinois, Chicago, Illinois
  - Translational Clinic of Corneal Neurobiology Laboratory, Illinois Eye and Ear Infirmary, University of Illinois, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tibrewal S, Sarkar J, Jassim SH, Gandhi S, Sonawane S, Chaudhary S, Byun YS, Ivanir Y, Hallak J, Horner JH, Newcomb M, Jain S. Tear fluid extracellular DNA: diagnostic and therapeutic implications in dry eye disease. Invest Ophthalmol Vis Sci. 2013 Dec 11;54(13):8051-61. doi: 10.1167/iovs.13-12844. PMID 24255046
- [Background] Sonawane S, Khanolkar V, Namavari A, Chaudhary S, Gandhi S, Tibrewal S, Jassim SH, Shaheen B, Hallak J, Horner JH, Newcomb M, Sarkar J, Jain S. Ocular surface extracellular DNA and nuclease activity imbalance: a new paradigm for inflammation in dry eye disease. Invest Ophthalmol Vis Sci. 2012 Dec 17;53(13):8253-63. doi: 10.1167/iovs.12-10430. PMID 23169882
- See also: Principal Investigator description — http://chicago.medicine.uic.edu/directory/name/sandeep-jain-md-jain/
- See also: Dry Eye and ocular GVHD Clinic at University of Illinois at Chicago — http://eyecare.uic.edu/clinics/DryEyeandOcularGVHDclinic.shtml
- See also: Corneal Neurobiology Laboratory (National Eye Institute funded) — http://cornealneurobiology.uic.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the clinical practice of the investigator at the time of their routine eye examination visit. The clinical practice is located in the Illinois Eye and Ear Infirmary (EEI), the University of Illinois at Chicago (UIC). The first participant was enrolled in May 2016, and the last participant was enrolled in February 2017.
Period: Overall Study
Arm/Group | Brimonidine 0.15% | Brimonidine 0.075% | Placebo
Started | 4 | 5 | 6
Completed | 3 | 2 | 5
Not Completed | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brimonidine 0.15% | Brimonidine 0.075% | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 6 | 13
  >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 3 | 3 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 4 | 5 | 5 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 6 | 15
Ocular Surface Disease Index (OSDI) [Mean (Standard Deviation); unit: units on a scale] — Ocular Surface Disease Index (OSDI), 12-item questionnaire, assesses symptom of ocular irritation in dry eye disease (DED) and how it affects functioning related to vision in past week. It has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on 0 to 4 scale with 0 being "none of the time" and 4 being "all of the time." OSDI score range from 0-100 with score 0-12 being normal, 13-22 being mild DED, 23-32 being moderate DED, and >33 being severe DED. OSDI=[(sum of scores for questions answered)×100]/[(total questions answered)×4]
  units on a scale | 48.4 (8.32) | 61.36 (22.42) | 56.03 (22.99) | 55.72 (20.28)
Schirmer I Test [Mean (Standard Deviation); unit: mm] — The Schirmer's I tests consists of a thin strip of filter paper placed in lower conjunctival fornix (between the lower eyelid and ocular surface) for 5 minutes. The length of wetting of the strip is used as a measure of tear production by the eye. A normal level of production is considered to be over 10 millimeters (mm) of tears on the paper. Anything under 10 mm is considered to be an abnormally low level of tear production. A measurement of less than 5 mm is considered severe dry eye.
  mm | 6.75 (8.42) | 2 (4.47) | 0.33 (0.74) | 1.4 (2.60)

OUTCOME MEASURES:

1. Primary Outcome: Primary Tolerability End Point: The Test Substance Tolerance (Visual Analog Scale) at 12 Weeks.
Description: Subjects assessed their tolerance to the administration of the study drug, utilizing a Visual Analog Scale (VAS). The VAS is a 100 mm horizontal line with verbal descriptors at either end and marks at an equal distance starting from 0 mm and leading up to 100 mm (0 10 20 30 40 50 60 70 80 90 100). The VAS ratings will be completed after administration of the study drug on Day 1 (post-dose), week 3, week 6, week 9 and week 12. Subjects will place a single slash mark across the horizontal line between the end labeled "completely intolerable" (0 mm) and "easily tolerable" (100mm).
Time Frame: 12 weeks
Population: The sponsor terminated the research early citing slow accrual of subjects and ceased sponsorship. At this point, the available valid sample size was 11 subjects at 12 weeks for assessing the tolerability at 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Brimonidine 0.15% | Brimonidine 0.075% | Placebo
Number analyzed (Participants) | 3 | 2 | 6
Participants
  Tolerability (100%) | 3 | 1 | 4
  Tolerability (95%) | 0 | 0 | 1
  Tolerability (90%) | 0 | 1 | 1
Statistical Analysis 1: Comparison: Brimonidine 0.15% vs Brimonidine 0.075% vs Placebo; We evaluated if the categorical type of tolerability measure is different between control (Artificial Tears) and intervention (Brimonidine, including both 0.15% high and 0.075% low doses groups); Test type: Other; p = 1, Fisher Exact; The type I error was adjusted by using the alpha spending function approach with O'Brien-Fleming type boundaries

ADVERSE EVENTS:
Time Frame: 4 months.
Arm/Group | Brimonidine 0.15% | Brimonidine 0.075% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/6

LIMITATIONS AND CAVEATS:
Given the inadequate power to detect efficacy (due to 40% enrollment), we did not perform an analysis to determine whether the drug had any beneficial effect. Due to slow accrual of subjects in this clinical trial sponsor ceased sponsorship.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT02975557/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT02975557/ICF_001.pdf